CLINICAL TRIAL: NCT02730637
Title: Prevention of Acute Kidney Injury Through Biomarker-guided Nephrological
Brief Title: Prevention of Acute Kidney Injury Through Biomarker-guided Nephrological Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Medical Center (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Kimmel, MD, MD, Robert Bosch Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RBK-348
Record Dates: First submitted 2016-03-18; First posted 2016-04-06 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

ARMS (2):
- Standard care (No Intervention): Patients with elevated biomarkers receive a standard treatment.
- Interventional care (Active Comparator): Patients in the interventional population receive an early nephrologist consultation which deliberates with attending doctor on preventing measures according to AKI-KDIGO recommendations.
  Interventions: Other: Early nephrologist consultation

INTERVENTIONS:
Other: Early nephrologist consultation
  Arms: Interventional care

SUMMARY:
This study examines the clinical relevance of early biomarkers to detect and prevent acute kidney injury. High-risk patients for developing acute kidney injury will be screened at initial presentation (emergency department and intensive care unit) for TIMP2xIGFBP7. In case of elevated readings patients will be randomized in two arms: The control group will be treated with standard care, the intervention group will receive an early nephrologic consultation.

DETAILED DESCRIPTION:
This study examines the impact of an early biomarker-guided intervention on the development of acute kidney injury (AKI). New biomarkers indicate kidney damage in an early stage before developing acute kidney injury according to AKI Kidney Disease Improving Global Outcomes (KDIGO) Definition is detectable. The investigators want to test if it's possible to prevent AKI based on elevated urinary biomarkers. Eligible patients will be randomly assigned to two groups, a control and an intervention Group by an early nephrologic consultation. The interventional group will receive an early preventive nephrologist consultation additionally to standard care.

ELIGIBILITY:
Inclusion Criteria:

* no acute kidney injury stage II-III (according to AKI KDIGO definition)
* urinary biomarker levels above cut-off
* inpatient treatment
* age ≥18 years
* informed consent or presumed will

Exclusion Criteria:

* existing acute kidney injury stage II-III (according to AKI KDIGO definition)
* age < 18 years
* end stage renal disease (ESRD), existing renal replacement therapy
* pregnancy
* withdrawal of consent
* missing presumed will

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI in both groups according to AKI KDIGO definition | within 24 hours

SECONDARY OUTCOMES:
Need for renal replacement therapy | within 24 hours
Need for renal replacement therapy | within 72 hours
Need for renal replacement therapy | within 30 days
Need for renal replacement therapy | within 60 days
Length of hospital stay | within 30 days
Length of hospital stay | within 60 days
Death | within 30 days
Death | within 60 days
Incidence of AKI in both groups according to AKI KDIGO definition | within 72 hours
Severety of AKI in both groups according to AKI KDIGO definition | within 72 hours
Incidence of AKI in both groups according to AKI KDIGO definition | within 30 days
Severity of AKI in both groups according to AKI KDIGO definition | within 30 days
Incidence of AKI in both groups according to AKI KDIGO definition | within 60 days
Severity of AKI in both groups according to AKI KDIGO definition | within 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kimmel, MD, Principal Investigator — Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF); Mark Dominik Alscher, MD, Principal Investigator — Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Locations (1):
- Robert-Bosch Hospital, Stuttgart, Germany

REFERENCES:
- [Derived] Schanz M, Wasser C, Allgaeuer S, Schricker S, Dippon J, Alscher MD, Kimmel M. Urinary [TIMP-2].[IGFBP7]-guided randomized controlled intervention trial to prevent acute kidney injury in the emergency department. Nephrol Dial Transplant. 2019 Nov 1;34(11):1902-1909. doi: 10.1093/ndt/gfy186. PMID 29961888